CLINICAL TRIAL: NCT06485583
Title: Comparison Between the Efficacy of CIMT and NDT Along With Conventional Physiotherapy Treatment on Upper Extremity Rehabilitation Among Patients of Stroke
Acronym: CIMT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shalamar Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, ayesha fatima, Principal Investigator, Shalamar Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ShalamarIHR
Record Dates: First submitted 2024-06-25; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Strokes Thrombotic
Keywords: (CIMT); (NDT)
MeSH Terms: conditions — Thrombotic Stroke | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Constraint-Induced Movement Therapy (Other): The rehabilitation plan involves several components to promote the recovery of the affected limb. Initially, we will immobilize the unaffected limb using a constraint device such as a mitt or sling for about 90% of waking hours over a period of six weeks.
  Interventions: Other: Constraint-induced movement therapy
- neurodevelopmental treatment (Other): The rehabilitation approach includes hands-on techniques to guide the patient through normal movement patterns. By providing sensory input, we aim to improve motor control and postural alignment, using techniques such as handling, guiding, and assisting movements.
  Interventions: Other: Neurodevelopmental Treatment

INTERVENTIONS:
Other: Constraint-induced movement therapy — is a rehabilitation technique used to improve motor function in people who have had a stroke or other neurological conditions. CIMT restricts the use of the unaffected limb, typically with a mitt or sling, to encourage the use of the affected limb.
  Arms: Constraint-Induced Movement Therapy
Other: Neurodevelopmental Treatment — Therapy, is a rehabilitation approach used to address movement and motor control deficits in people with neurological illnesses such as stroke, cerebral palsy, or traumatic brain injury.
  Arms: neurodevelopmental treatment

SUMMARY:
To compare the efficacy of CIMT and NDT among stroke patients To study the phenomena of transfer of training To study relationship between the MMSE score and stroke rehabilitation

DETAILED DESCRIPTION:
This research aims to provide a comprehensive comparison of CIMT and NDT, supplemented by conventional physiotherapy, in the rehabilitation of upper extremity function among stroke patients. The findings will inform clinical practice, guiding the development of optimized, patient-centered rehabilitation strategies.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be aged 40-65 years and will have experienced either a hemorrhagic or ischemic stroke with hemiplegic presentation within the past 1 to 6 months. Additionally, they must have a Mini-Mental State Examination (MMSE) score of 23.

Exclusion Criteria:

* Participants with visual or auditory deficits, musculoskeletal (MSK) disorders, mental impairments, or a history of surgery will be excluded from the study.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-06-28 (Estimated); Primary Completion 2024-11-29 (Estimated); Study Completion 2025-01-29 (Estimated)

PRIMARY OUTCOMES:
upper extremity rehabilitation | 6 WEEKS
  The Motor Assessment Scale (MAS) by Carr and Shepherd is a clinical tool used to evaluate upper extremity rehabilitation in stroke patients. It assesses motor recovery through eight items, each reflecting daily activities, scored on a 7-point scale from 0 (unable to perform) to 6 (optimal performance). For upper extremity assessment, the MAS includes tasks like hand movements (grasping, releasing, manipulating objects), advanced hand activities (fine motor skills such as writing or buttoning a shirt), and upper arm function (reaching, lifting, placing objects). Patients perform these tasks while clinicians observe and score their performance. The MAS provides a quantitative measure of motor recovery, facilitating progress tracking, goal setting, and personalized therapy interventions, making it a reliable and straightforward tool for capturing functional changes in stroke patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Ayesha Fatima, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Kwakkel G, Veerbeek JM, van Wegen EE, Wolf SL. Constraint-induced movement therapy after stroke. The Lancet Neurology. 201514(2):224-34. 2. Uswatte G, Taub E. Constraint-induced movement therapy: a method for harnessing neuroplasticity to Page 5 of 7 treat motor disorders. Progress in brain research. 2013207:379-401. 3. Budhota A, Chua KSG, Hussain A, Kager S, Cherpin A, Contu S, et al. Robotic Assisted Upper Limb Training Post Stroke: A Randomized Control Trial Using Combinatory Approach Toward Reducing Workforce Demands. Frontiers in neurology. 202112:622014. 4. Folstein MF, Folstein SE, McHugh PR. Mini-mental state: A practical method for grading the cognitive state of patients for the clinician. Journal of Psychiatric Research. 197512(3):189-98. 5. Bohannon RW, Smith MB. Interrater reliability of a modified Ashworth scale of muscle spasticity. Phys Ther. 198767(2):206-7. 6. Carr JH, Shepherd RB, Nordholm L, Lynne D. Investigation of a new motor assessment scale for stroke patients. Phys Ther. 198565(2):175-80. 7. Ahn SY, Bok S-K, Lee JY, Ryoo HW, Lee HY, Park HJ, et al. Benefits of Robot-Assisted Upper-Limb Rehabilitation from the Subacute Stage after a Stroke of Varying Severity: A Multicenter Randomized Controlled Trial. Journal of Clinical Medicine. 202413(3):808. 8. Winstein CJ, Wolf SL, Dromerick AW, Lane CJ, Nelsen MA, Lewthwaite R, et al. Effect of a Task-Oriented Rehabilitation Program on Upper Extremity Recovery Following Motor Stroke: The ICARE Randomized Clinical Trial. JAMA. 2016315(6):571-81. 9. Sakzewski L, Ziviani J, Abbott DF, Macdonell RA, Jackson GD, Boyd RN. Randomized trial of constraint-induced movement therapy and bimanual training on activity outcomes for children with congenital hemiplegia. Developmental medicine and child neurology. 201153(4):313-20.